CLINICAL TRIAL: NCT04913883
Title: Adjustment of Astigmatism for Laser Correction Using Vector Planning Calculator
Brief Title: Laser Correction of Astigmatism Using Vector Analysis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Fathy Rateb Hassan, Resident Ophthalmologist at Assiut Police Hospital, Assiut University
Other Study IDs: Adjustment of Astigmatism
Record Dates: First submitted 2021-05-25; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine the effectiveness of correcting astigmatism by laser refractive surgery by a vectorial astigmatism outcome analysis that uses 3 fundamental vectors : target induced astigmatism vector ( TIA) , surgically induced astigmatism vector , and difference vector , as described by Alpins method.

DETAILED DESCRIPTION:
Astigmatism is a condition of the eye where the cornea (clear window in front of the eye) has 2 different curvatures (much like an American football cut in half) so that, instead of being a single focal point, there ends up being two different focal points, neither of which is in focus.

As you can imagine, this makes whatever you are looking at blurred and fuzzy like a camera out of focus. Both objects up close and far away can look blurred and fuzzy with astigmatism. Many people with astigmatism also are nearsighted or farsighted.

There are several different treatment options if you have astigmatism with or without nearsightedness or farsightedness. Various treatment options available from an eye specialist include: Glasses, Contact Lenses and Laser Eye Surgery

Laser Eye Surgery:

Laser eye surgery, or laser vision correction, involves using lasers to reshape the front surface (cornea) of your eyes so that you can focus better. It can correct short-sightedness , long-sightedness and astigmatism.There are several different laser eye surgery options that can be used to help correct vision problems caused by astigmatism.Laser eye surgery corrects the refractive error in the cornea so that, instead of there being two focal points, there will be only one focal point that is in focus post-surgery.Laser vision correction can be used if you have astigmatism with or without nearsightedness or farsightedness.However, what laser eye procedures you are an ideal candidate for will vary based on your vision correction needs LASIK( Laser ASsisted In-situ Keratomileusis ),PRK ( Photorefractive Keratectomy ) and SMILE (Small Incision Lenticule Extraction ) . Unlike glasses or contacts, which just address astigmatism so you can see clearly with assistive devices, laser eye surgery is the only treatment to potentially resolve astigmatism so you no longer need glasses or contacts. To determine the effectiveness of correcting astigmatism by laser refractive surgery by a vectorial astigmatism outcome analysis that uses 3 fundamental vectors: target induced astigmatism vector (TIAT), surgically induced astigmatism vector, and difference vector, as described by the Alpins method.

Alpins method :

This method of astigmatism analysis enables the examination of results of astigmatism treatment by both refractive and corneal measurements. The approach uses vector analysis, which is used in this series for examining regular astigmatism. This can be further applied to irregular astigmatism by separately examining the 2 halves of the cornea by adding a second analysis between 181and 360 degrees and displaying both together on a 360 degree polar diagram as they would appear on an eye or topography map drawn between the two points . The length of this line represents the WTW ( White To White ) value [16].

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age .
* Stable eyeglass and contact lenses prescription for at least 2 to 3 years .
* Stable vision over at least the past year .
* No history or findings of active corneal disease .
* No significant dry eye .
* Not pregnancy or nursing .
* Refractive cylinder more than -1D (Diopter) .

Exclusion Criteria:

Certain conditions make the method inadvisable :

* Residual , recurrent or active ocular disease such as uveitis , sever dry eyes , sever allergic eye disease , glaucoma visually significant cataract , and retinal disease .
* Previous corneal surgery or trauma within the corneal flap zone .
* Patent corneal vascularisation within 1mm of the corneal flap zone .
* Age less than 18 years old .
* Pregnancy or breast feeding .
* Certain medical conditions such as autoimmune diseases (eg. lupus , rheumatoid arthritis), immunodeficiency states (eg. HIV) and diabetes may prevent proper healing after a refractive procedure.
* Systemic medications likely to affect wound healing such as retinoic acid and steroids .
* Keratoconus or other active eye disease .

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: Study will include 50 patients in different ages .
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
. Post operative Visual Acuity | one year
  To determine the effectiveness of correcting astigmatism by laser refractive surgery by a vectorial astigmatism outcome analysis by : CDVA and UCDVA, pentacam , 3 month, 6 month and 1 year after surgery.
  * 3 months postoperative : assessment of visual acuity using corrected distance visual acuity (CDVA) , and uncorrected distance visual acuity (UCDVA) and pentacam measures .
  * 6 months postoperative : assessment of visual acuity using corrected distance visual acuity (CDVA) , and uncorrected distance visual acuity (UCDVA) and pentacam measures .
  * One year postoperative : assessment of visual acuity using corrected distance visual acuity (CDVA) , and uncorrected distance visual acuity (UCDVA) and pentacam measures .

SECONDARY OUTCOMES:
Postoperative Assessment | 3 months
  Wavefront Analysis of post operative corneal results , 3 months after surgery to assess visual acuity . wavefront analysis is that it measures the entire visual system, rather than just the corneal surface, as in corneal topography.

CONTACTS AND LOCATIONS:
Overall Officials: Abdelnasser Awad, Professor, Principal Investigator — Ophthalmology Department; Khaled Abdelazeem, Asst. Prof, Principal Investigator — Ophthalmology Department; Mohamed Anwer, Lecturer, Principal Investigator — Ophthalmology Department

REFERENCES:
- [Background] Alpins N. Astigmatism analysis by the Alpins method. J Cataract Refract Surg. 2001 Jan;27(1):31-49. doi: 10.1016/s0886-3350(00)00798-7. PMID 11165856